CLINICAL TRIAL: NCT02841371
Title: Early Screening and Diagnosis of Chronic Kidney Disease
Brief Title: Early Screening and Diagnosis of CKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ES-CKD
Record Dates: First submitted 2016-07-13; First posted 2016-07-22 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Kidney; Disease (Functional); Chronic Kidney Disease
Keywords: estimated glomerular filtration rate; serum creatinine; serum cystatin C; chronic kidney disease
MeSH Terms: conditions — Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- chronic kidney disease (CKD): chronic kidney disease (CKD) is defined as abnormalities of kidney structure (markers of kidney damage) or function (decreased GFR by 99mTc-DTPA renal clearance and/or eGFR), present for more than 3 months.
  Interventions: Radiation: 99mTc-DTPA
- no CKD: Suspected chronic kidney disease but no chronic kidney disease after screening by abnormalities of kidney structure (markers of kidney damage) or function (decreased GFR by 99mTc-DTPA renal clearance and/or eGFR), present for less than 3 months, or no abnormalities of kidney structure or function.
  Interventions: Radiation: 99mTc-DTPA

INTERVENTIONS:
Radiation: 99mTc-DTPA — a 99mTc-DTPA renal dynamic imaging measurement as the reference glomerular filtration rate (rGFR).
  Other Names: technetium-99m-labeled diethylenetriaminepentaacetic acid

SUMMARY:
Chronic kidney disease (CKD) is a global public health problem. The prevalence of CKD in adults in China was 10.8%. Albuminuria measurement and estimating glomerular filtration rate (GFR) are the primary means of screening for CKD in epidemiological investigations. However, there are many important problems to be solved, whether albuminuria test or GFR evaluation. The investigators aim to detect thrice albumin-creatinine ratio (ACR) within three months, with simultaneous test of urinary protein-creatinine ratio (PCR), 24-hour urine protein excretion rate (PER) and 24-hour albumin albumin excretion rate (AER) to compare the effects of different times of screening for CKD and observe the daily physiological variation of ACR, PCR, AER and PER, derive ACR and PCR reference value on the basis of different genders, in order to facilitate the early diagnosis of CKD. Meanwhile, for more accurate assessment of GFR in Chinese populations, the investigators intend to validate beta-trace protein (BTP) based equation to evaluate GFR compared with 99mTc-diethylenetriamine pentaacetic acid (DTPA) renal clearance method. Then to develop GFR estimation equation based on the combination of serum creatinine, cystatin C, β2 -microglobulin and BTP applicable in China.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a global public health problem. The prevalence of CKD in adults in China was 10.8%. Awareness of CKD is only 10.04% from a national cross-sectional survey in China. CKD is characterised by decreased estimated glomerular filtration rate (eGFR) and increased albuminuria, present for more than three months, and is associated with adverse outcomes (all-cause mortality, acute kidney injury, and end-stage renal disease), independent of hypertension and diabetes, age, or sex. CKD may carry a coronary heart disease risk similar to that of diabetes. The estimated lifetime risk of CKD stage 3a was more than 50%, lower than that of hypertension (83%-90% for a 55-year-old), but higher than those for diabetes (33%-39%), coronary heart disease (32%-49% for a 40-year-old), and invasive cancer (38%-45%).

Albuminuria measurement and estimating glomerular filtration rate (GFR) are the primary means of screening for CKD in epidemiological investigations. However, there are many important problems to be solved, whether albuminuria test or GFR evaluation. The investigators aim to detect thrice albumin-creatinine ratio (ACR) within three months, with simultaneous test of urinary protein-creatinine ratio (PCR), 24-hour urine protein excretion rate (PER) and 24-hour albumin excretion rate (AER) to compare the effects of different times of screening for CKD and observe the daily physiological variation of ACR, PCR, AER and PER, and repeat test to reduce the physiological variation, and further derive ACR and PCR reference value on the basis of different genders, in order to facilitate the early diagnosis of CKD. Meanwhile, for more accurate assessment of GFR in Chinese populations, the investigators intend to validate beta-trace protein (BTP) based equation to evaluate GFR compared with 99mTc-diethylenetriamine pentaacetic acid (DTPA) renal clearance method. Then the investigators aim to develop GFR estimation equation based on the combination of serum creatinine, cystatin C, β2-microglobulin and BTP applicable in China, for early and accurate assessment of GFR in Chinese people, and develop appropriate software to estimating GFR.

ELIGIBILITY:
Inclusion Criteria:

* Health examination population at the department of nephrology
* Chronic kidney disease

Exclusion Criteria:

* Severe heart failure
* Acute renal failure
* Pleural or abdominal effusion
* Serious edema or malnutrition
* Skeletal muscle atrophy
* Amputation
* Ketoacidosis
* Patients who were taking trimethoprim or cimetidine or angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blocker (ARB)
* Patients who had recently received glucocorticoid and hemodialysis therapy
* Female during the menstrual period
* Pregnant woman
* Who unable to sign informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese participants with CKD were selected from Nanjing First Hospital in China. All patients met the diagnostic criteria of CKD according to National Kidney Foundation-Kidney Disease Outcomes Quality Initiative (K/DOQI) clinical practice guidelines.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bias of estimated GFR less than 5 ml per minute per 1.73 m2 versus reference GFR | 1 year
  Bias was defined as the median results of differences between estimated GFR and reference GFR (eGFR- rGFR).
Precision of estimated GFR less than 30 ml per minute per 1.73 m2 versus reference GFR | 1 year
  Precision was defined as the interquartile range (IQR) of the differences between estimated GFR and reference GFR.
Accuracy of estimated GFR more than 70% | 1 year
  Accuracy was calculated as the proportion of estimated GFR within 30% of reference GFR.

SECONDARY OUTCOMES:
net reclassification index more than 10% | 1 year
  Net reclassification improvement (NRI) was defined as the sum of those classified upward to higher risk in those with an event plus those classified downward to lower risk in those without an event less the sum of those classified downward to lower risk in those with an event plus those classified to higher risk in those without an event. The event in this study was having a measured GFR that was less than 60 ml per minute per 1.73 m2.
Composite outcomes of sensitivity of a single screen using estimated GFR and/or albuminuria to detect CKD more than 0.6, or specificity of a single screen using estimated GFR and/or albuminuria to detect CKD more than 0.8 | 1 year
  Sensitivity of a single screen using estimated GFR and/or albuminuria to detect CKD more than 0.6, or specificity of a single screen using estimated GFR and/or albuminuria to detect CKD more than 0.8

CONTACTS AND LOCATIONS:
Overall Officials: Xin Du, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided